CLINICAL TRIAL: NCT00315666
Title: Prophylactic Effect of Memantine in Chronic Tension-Type Headache
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Danish Headache Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2006-000060-82; KA-20060021
Record Dates: First submitted 2006-04-18; First posted 2006-04-19 (Estimated); Last update posted 2009-02-20 (Estimated); Status verified 2009-02

CONDITIONS: Tension-Type Headache
Keywords: Chronic tension-type headache
MeSH Terms: conditions — Tension-Type Headache | interventions — Memantine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: memantine

SUMMARY:
The purpose of this study is to test whether memantine has a prophylactic effect on chronic tension-type headaches.

ELIGIBILITY:
Inclusion Criteria:

* Chronic tension-type headache
* Normal urine pH

Exclusion Criteria:

* More than 1 migraine attack/month
* Other major illnesses
* Overuse of medicine/alcohol
* Women not using AC
* Pregnant/breast-feeding women
* Allergy to memantine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2006-05; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Headache duration
Headache intensity

SECONDARY OUTCOMES:
Headache frequency
The use of simple analgesics
Side effects

CONTACTS AND LOCATIONS:
Overall Officials: Lars Bendtsen, MD, PhD, Principal Investigator — Danish Headaches Center, Dept. of Neurology, KAS Glostrup, DK-2600 Glostrup
Locations (1):
- Danish Headaches Center, Glostrup Municipality, Denmark